CLINICAL TRIAL: NCT02190227
Title: Tumor RNA Disruption Assay as a Tool to Predict Response to Neoadjuvant Chemotherapy in Breast Cancer: Optimizing Timing of Biopsy
Brief Title: RNA Disruption Assay (RDA) Response Prediction in Neoadjuvant Chemotherapy Breast Cancer Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Laurentian University (Other)
Responsible Party: Principal Investigator, Jean-Fancois Boileau, Surgical Oncologist and Clinician-Researcher, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MJGH-RDA
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Invasive Breast Cancer
Keywords: Breast Cancer; Chemotherapy; Neoadjuvant; RNA Disruption Assay; Biopsies; Response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tumor RDA biopsy (Other): Tumor RDA score measured from an FNA biopsy after cycle 1-2-3 of neoadjuvant chemotherapy and after first cycle of second chemotherapy agent if palpable tumour present.
  Interventions: Device: Tumor RDA biopsy

INTERVENTIONS:
Device: Tumor RDA biopsy — Tumor RDA score measured from an FNA biopsy after cycle 1-2-3 of neoadjuvant chemotherapy and after first cycle of second chemotherapy agent if palpable tumour present.

SUMMARY:
The purpose of this study is to determine the optimal time to use the Tumor RNA Disruption Assay (RDA) as a predictor of pathological complete response (pCR) in patients with breast cancer treated with neoadjuvant chemotherapy.

This is important because the earlier non-responders are identified, the greater is the impact of reducing side effects of ineffective treatments.

The study hypothesis is that the RDA score will accurately predict for tumor response after one cycle of chemotherapy.

DETAILED DESCRIPTION:
This prospective clinical trial will determine if the tumor RDA score can predict for pCR after the first, second, and third cycles of chemotherapy in women with breast cancer treated with neoadjuvant therapy. Tumor RDA score will also be measured after the first dose of any new chemotherapy agent if residual palpable disease is present.

Data will be collected until accrual target of 30 patients is met. All patients will undergo core needle biopsy of the breast tumor and analysis of ER, PR, and HER-2-Neu receptors. Patients will receive neoadjuvant therapy as recommended by their treating physicians. All chemotherapy regimens will be acceptable for participation in this study. Usually, these regimens are between 6 to 8 cycles, often with a switch of chemotherapy regimens after 3 to 4 cycles.

Evaluation of tumor size will be determined by 2 axis tumor measurement performed prior to, and after each chemotherapy treatment. The Tumor RDA score will be evaluated by performing fine needle aspiration (FNA) biopsies under local anesthetic, if the tumor is clinically palpable, after the first, second, and third cycles of chemotherapy. Tumor RDA score will also be determined if palpable tumor is present after the first cycle of any second chemotherapy agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female.
* Patients must be 18 years of age or older.
* Patients with stage I, II, or III breast cancer that is greater or equal to 2 cm on clinical examination.
* Patients that have biopsy proven invasive breast cancer diagnosed by core needle biopsy
* Patients who are chemotherapy and radiotherapy naïve for the treatment of the current breast cancer.
* Patients that accept to undergo neoadjuvant chemotherapy.
* Patients with bilateral breast cancer are eligible.
* Patients that understand, accept, and have signed the approved written consent form.
* Patients will need to consent to be part of the study.

Exclusion Criteria:

Patients with one or more of the following conditions are ineligible for this study:

* Patients who have had previous surgery, chemotherapy or radiotherapy for the current breast cancer
* Patients who are pregnant or breast feeding.
* Psychiatric or addictive disorders or conditions or social factors that may preclude the patient from meeting study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR). | At time of surgery (4-8 months after first dose of neoadjuvant therapy).
  Determine the optimal time at which Tumor RNA Disruption Assay (RDA) can predict pathological complete response (pCR) in patients with breast cancer treated with neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Boileau, MD MSc FRCSC, Principal Investigator — McGill University, Montreal, Quebec, Canada
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Parissenti AM, Chapman JA, Kahn HJ, Guo B, Han L, O'Brien P, Clemons MP, Jong R, Dent R, Fitzgerald B, Pritchard KI, Shepherd LE, Trudeau ME. Association of low tumor RNA integrity with response to chemotherapy in breast cancer patients. Breast Cancer Res Treat. 2010 Jan;119(2):347-56. doi: 10.1007/s10549-009-0531-x. PMID 19771508